CLINICAL TRIAL: NCT07293468
Title: Comparison of Stereotactic Body Radiotherapy and Selective Internal Radiation Therapy in Combination With Immunotherapy for Locally-advanced, Unresectable Hepatocellular Carcinomas: an Open-label, Randomized Controlled Trial (BIIRTH)
Brief Title: Comparison of SBRT and SIRT With Combination IO for Locally-advanced, Unresectable HCCs (BIIRTH)
Acronym: BIIRTH
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Collaborators: Queen Mary Hospital, Hong Kong (Other); The University of Hong Kong (Other); The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Wong Sean Man Natalie, Principal Investigator, Tuen Mun Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIIRTH
Record Dates: First submitted 2024-12-05; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: TACE; SBRT; Y90; SIRT; immunotherapy; combination therapy; locally advanced; unresectable HCC; RCT; liver; hepatocellular carcinoma; stereotactic body radiotherapy; transarterial chemoembolization; radioembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; atezolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: This is an investigator-initiated, phase III, prospective, open-label, multi-institutional randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TACE-SBRT arm (Experimental): Combination TACE and SBRT followed by immunotherapy
  Interventions: Procedure: Transarterial chemoembolization (TACE); Radiation: Stereotactic Body Radiation Therapy (SBRT); Drug: Atezolizumab & Bevacizumab
- Y90 SIRT arm (Active Comparator): Combination Y90 SIRT followed by immunotherapy
  Interventions: Radiation: SIRT Yttrium-90; Drug: Atezolizumab & Bevacizumab

INTERVENTIONS:
Procedure: Transarterial chemoembolization (TACE) — One dose of TACE would be performed as per standardized procedure at 21-35 days preceding SBRT. Celiac and superior mesenteric arterial and porto-venogram would be performed to exclude main portal vein occlusion and to delineate the size(s) and number(s) of tumour nodule(s). Supra-selective cannulation of the supplying tumour artery would follow. The 1:1 lipiodol-cisplatin emulsion prepared by pumping would be slowly injected under fluoroscopic guidance according to the tumour size and arterial blood flow.
  Arms: TACE-SBRT arm
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Patients are immobilized with customized device and abdominal compression or active breathing control. Four-dimensional computed tomography (4D-CT) was phase-sorted into 10 image-sets. A radiation dose of 27.5-50.0 Gy in five fractions, delivered in alternate days, is allowed. The prescription dose is individualized based on normal tissue constraints. This should be based on delivering a maximal tumoricidal dose while respecting the tolerance dose of neighbouring organs-at-risk. SBRT is delivered by dynamic conformal arc therapy, intensity-modulated RT, or volumetric modulated arc RT.
  Arms: TACE-SBRT arm
Radiation: SIRT Yttrium-90 — Patients undergo intrahepatic arterial Y90-radioembolisation (TheraSphere glass microspheres; MDS Nordion, Ottawa, Canada or SIR-Spheres, Sirtex Medical Pty Limited; St. Leonards, NSW, Australia). The administered activity of Y90-glass microspheres was determined by the nuclear medicine physician, medical physicist, radiologist and clinical oncologist using the artery-specific partition model within the limits of radiation safety, taking into account treatment variables including patient's body surface area, tumour-to-normal liver ratio, and liver tumour size. Where possible, personalized dosimetry using the partition model was the default methodology to facilitate selective administration of Y90-radioembolisation avoiding toxicities to the normal liver parenchyma.
  Arms: Y90 SIRT arm
Drug: Atezolizumab & Bevacizumab — Patients will start Atezolizumab-bevacizumab 14days upon completion of SBRT or SIRT. Atezolizumab, if given, is administered via IV infusion at a fixed dose of 1200mg, together with Bevacizumab (start 28days after SBRT/SIRT) via IV infusion at a fixed dose of 15mg/kg, on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator, or after curative surgical intervention is performed with no evidence of residual disease. Patients who transiently or permanently discontinued either atezolizumab or bevacizumab due to an adverse event are allowed to continue with single-agent therapy provided there is ongoing clinical benefit as determined by the investigator.

SUMMARY:
The goal of this clinical trial is to compare the safety and efficacy of sequential Transarterial Chemoembolization (TACE) and Stereotactic body radiation therapy (SBRT) versus Y90-radioembolisation (SIRT), followed by systemic therapy in patients with large, locally advanced, unresectable Hepatocellular carcinoma (HCC).

The main question it aims to answer is whether Sequential TACE-SBRT potentially gives longer Progression-free survival (PFS) benefit with similar toxicities as compared with Y90 SIRT.

Participants will be recruited via multidisciplinary meetings (MDTs) with hepatobiliary surgeons, medical hepatologists and radiologists with consistent, strict considerations on eligibility and treatment alternatives. Eligible patients will be randomized in 1:1 ratio to received one of the two treatment arms.

DETAILED DESCRIPTION:
1. Background

Hepatocellular carcinoma (HCC) represents a major global health threat, ranking sixth in worldwide cancer incidence and third in cancer mortalities.(1) Southeast Asia remains endemic, with liver cancer ranking fifth and third in local cancer incidence and mortalities respectively according to the Hong Kong Cancer Registry.(2) While resection, radiofrequency ablation (RFA) and liver transplantation represents chances of cure, only 30% of patients are eligible for curative local intervention upon presentation. Large, locally advanced HCCs represent a distinct population of aggressive clinical courses conferring poor prognoses and are often rapidly symptomatic, with limited treatment options and represent true unmet clinical needs.(3)

1.1 Current Landscape of Locoregional Therapies for Locally Advanced HCC A substantial population of locally advanced HCC patients die of intra-hepatic treatment failures. Intensifying local treatment strategies has been suggested to improve survival outcomes, hence optimizing locoregional therapy is of paramount importance.(4) Transarterial chemoembolization (TACE) remains the most widely adopted local treatment modality in unresectable HCCs. Growing evidence, however, has demonstrated limited efficacy among large tumours, with reported low response rates of roughly 30% among large (≥5cm) or multinodular HCCs and poor 2-year overall survival of 0% for tumour sizes ≥8 cm.(5)

On the other hand, radiotherapy techniques have evolved, with stereotactic body radiotherapy (SBRT) and selective internal radiotherapy (SIRT) gaining recognition in the treatment of large unresectable HCCs.(6) SIRT has been suggested to be as effective as sorafenib in HCC patients with liver-only involvement with more favourable tumour response and side effect profile. Lately, the American Society for Radiation Oncology (ASTRO) Clinical Practice Guideline on External Beam Radiotherapy (EBRT) for Primary Liver Cancers 2021 recommended EBRT as a potential first-line therapy option in liver-confined, incurable HCCs alongside with catheter-based therapies including TACE and SIRT.(7)

While Y90 SIRT is considered the Hospital Authority's standard in HCC patients with tumours (i) ≥8cm, or (ii) presence of portal vein invasion, or (iii) as a bridge therapy to liver transplantation(8), there is currently no prospective, head-to-head comparison on the choice of locoregional therapy, and growing evidence urges optimization and standardization of treatment algorithms for locally advanced, unresectable tumours.

1.1.1 SIRT Radioembolization with 90yttrium (Y90)-tagged glass or resin microspheres has been an internationally recognized and widely-practiced local treatment modality among large, unresectable HCCs. Salem et al reported comparable outcomes to TACE in terms of response rate (42%) and time-to-progression (7.9 months) for a sample of 291 patients with median tumour sizes of 7 cm with acceptable toxicities.(9) As Hospital Authority's standard indication, Y90 SIRT is considered in HCC patients with tumours (i) ≥8cm, or (ii) presence of portal vein invasion, or (iii) as a bridge therapy to liver transplantation.(8)

However, price and accessibility concerns have limited its application, especially among pandemic areas and/or developing countries. In addition, more vigorous screening is required to meet the eligibility criteria for SIRT. In particular, a pre-treatment Technetium-99m (99mTc) macroaggregated albumin (MAA) scan is required as initial screening, in which only patients without significant lung shunting of hepatic artery blood flow are considered eligible. While HCC patients were found to have higher median lung shunt fraction (LSF) than other metastatic liver tumours, as high as 21.4% were ineligible for Y90 due to an exceedingly high LSF.(10)

1.1.2 TACE with SBRT SBRT liver has emerged as a promising local therapy in patients with locally advanced HCCs. While TACE alone might be suboptimal in treating large, unresectable HCCs, meta-analyses concluded an improvement in OS with combination TACE and EBRT as compared to TACE alone.(11) Furthermore, a retrospective study of patients with unresectable HCCs and a median tumour size of 8.5cm (5.1-21cm) demonstrated a significantly better 5-year OS rate of 46.9% vs 32.9% among those who received combination TACE and SBRT versus SBRT alone.(12)

The American Society for Radiation Oncology (ASTRO) clinical practice guideline on EBRT for primary liver cancers conditionally recommended the use of EBRT in patients with liver-confined, multifocal and/or unresectable HCCs, with or without macrovascular invasion, either alone or sequenced with other catheter-based therapies.(7) The relatively high accessibility, less expensive RT and TACE interventional radiology facilities has represented a highly attractive treatment option.

Prior local work has been done. A substantially enhanced anti-tumour response and survival benefits with similar toxicities by means of sequential single-course of TACE followed by SBRT as compared with the TACE alone group by propensity score matched analysis was reported.(13) Subsequently, a published 2020 study evaluating 55 consecutive patients with large (≥10 cm) HCCs of median tumour sizes 15.3cm (range, 10.0-25.7cm) receiving sequential TACE and hypofractionated image-guided radiotherapy (HIGRT) at Tuen Mun Hospital during 2007-2017 with a 1-year local in-field progression-free survival (PFS) rate of 57.4% (95% CI = 40.8%-74.0%). Notably, 27% of treatment responders achieved remarkable tumour downstaging and underwent subsequent curative resection, achieving a significantly prolonged OS of 41.2months (95% CI, 19.1-63.2 months) as compared to those without surgery. (14) Such results are also in line with the Hong Kong consensus statements on unresectable HCC 2021 guidelines affirming the role of combination TACE and SBRT.(15)

1.1.3 Immune Checkpoint Inhibitors (ICI) While systemic therapy is also considered a standard therapeutic option in locally advanced, unresectable HCCs,(16) response rates were modest even in the post-immunotherapy era, ranging from 5-40%.(17,18) Atezolizumab, a programmed death ligand 1 (PD-L1) inhibitor, in combination with bevacizumab, a monoclonal antibody against the vascular endothelial growth factor (VEGF), is the preferred first-line treatment option since the establishment of IMbrave150 trial.(18) The response rate at 27.3% (95% CI, 7.4-18.0%), albeit the presence of survival benefits, urges needs for further improvement.(18)

1.2 Emerging Combination of Locoregional and Systemic Therapy and Potential Surgical Conversion in Local Advanced HCCs

Evolving evidence suggests upfront liver-directed therapy application followed by systemic therapy combination could achieve successful tumour downstaging in locally advanced HCCs leading to curative surgeries and improved survival. The randomized, multicentre, phase 3 NRG/RTOG 1112 trial reported the addition of SBRT to sorafenib has improved OS, PFS and TTP in advanced HCC patients versus Sorafenib alone, with no significant increase in adverse events.(19) Another recent prospective single arm, single centre, phase 2 NASIR-HCC study demonstrated rates of surgical conversion (9.5%), partial response (PR) (16.7%) and OR (41.5%; 95% CI: 26.3-57.9%), as well as median time to progression (mTTP) of 8.8months (95% CI: 7.0-10.5months) and mOS of 20.9months (95% CI: 17.7-24.1months) in 42patients with HCCs exceeding 5cm or multiple beyond the up-to-seven criteria treated with SIRT followed by nivolumab combination therapy.(20)

Moreover, local research is emerging. The published START-FIT study in Lancet Gastroenterology and Hepatology was a prospective single arm, multi-centre phase 2 trial demonstrating initial success of the novel, sequential TACE-SBRT-immunotherapy (avelumab) approach. Promising rates of conversion (55%), complete response (CR) (42%) and objective response (OR) (66.7%; 95% CI: 48.2-82.0%), as well as favourable mPFS of 20.7months (95% CI: 14.6-26.8months) and median overall survival (mOS) of 30.3months (95% CI: 22.7-37.8months) were achieved in 33 patients with locally advanced, upfront unresectable HCCs of median sizes 15.1cm (range: 5.3-31.1cm). Toxicity profile was also favourable, hereby demonstrating the safety and efficacy of our combination TACE-SBRT and immunotherapy treatment. (21) Since then, two propensity score matching analyses, one of which was in Liver Cancer, demonstrated a significantly improved OS rates of SBRT-immunotherapy as compared to TACE alone (2-year OS 80.4% vs. 8.3%), and SBRT alone (3-year OS 62.9% vs. 43.4%) respectively. (22,23)

While sequential local-systemic therapy is expected to be synergistic, direct comparison on the different types of local therapy backbone is lacking. Determining the optimal loco-systemic treatment strategy is therefore integral to achieve potential surgical conversion and unlock major survival benefits.

With results of combination TACE and SBRT being numerically favourable as compared to that of SIRT, a comparison of sequential TACE-SBRT versus Y90 SIRT would therefore be the next logical investigation approach. We aim at conducting a prospective trial with head-to-head comparison on combinational TACE-SBRT versus Y90 SIRT as standard locoregional therapy, together with combination immunotherapy treatment among locally advanced HCCs.

This project carries substantial impact on HCC management via (1) establishing the role of locoregional therapy in the post-immunotherapy era, (2) shedding light on local and international guidelines of incorporating locoregional therapy to first-line treatment in locally advanced HCC patients, and (3) potentially unlocking major, durable survival benefits through the synergistic effects of optimal local-systemic therapy combination among patients with locally advanced HCCs whom prognosis is guarded and treatment option is limited.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with HCC either by histology or by the American Association for the Study of Liver Diseases Criteria (AASLD) 2018
* Patients age 18-80 years of age with HCCs deemed unresectable at the Multidisciplinary Team Meetings (MDTs) because of the following:
* R0 resection not feasible e.g. unfavourable tumour location
* Remnant liver volume <30% in non-cirrhotic patients or 40% in cirrhotic patients
* Indocyanine green test >15%
* Patients with Barcelona Clinic Liver Cancer (BCLC) stage B2-4 (unresectable group) or C
* Tumour sizes of ≥5cm, of which ≥1 is a measurable lesion as defined by the mRECIST criteria
* Subjects aged 18-80 years of age
* ECOG performance status of 0-1
* Predicted life expectancy should be of ≥ 3 months
* Child Pugh (CP) score of A5-B7
* Adequate organ and marrow functions, as listed below:
* Haemoglobin ≥9 g/dL
* Absolute neutrophil count ≥1,500/uL
* Platelet count ≥100,000/L
* Total bilirubin ≤2.0 x upper limit of normal (ULN)
* Albumin ≥2.8 g/dL
* ALT ≤3 x ULN
* INR ≤1.6
* Calculated creatinine clearance (eGFR) ≥45 mL/minute as determined by Cockcroft-Gault (using actual body weight) or 24-hour urine creatinine clearance
* Liver volume minus intrahepatic gross tumour volume (GTV) with >700cc
* Patients with concomitant HBV infection (defined as having HBsAg positive and/or detectable HBV DNA level) must be treated with antiviral therapy (per local institutional practice) to ensure adequate viral suppression (defined as HBV DNA <2,000 IU/mL) prior to enrolment, throughout study duration and continue for at least 6 months following the last dose of local-systemic therapy
* Informed consent provided
* Females of childbearing potential or non-sterilized male who are sexually active must use a highly effective method of contraception
* Females of childbearing potential must have negative serum or urine pregnancy test

Exclusion Criteria:

* Prior invasive malignancy within 2 years except for noninvasive malignancies such as cervical carcinoma in situ, in situ prostate cancer, non-melanomatous carcinoma of the skin, lobular or ductal carcinoma in situ of the breast that has been surgically cured
* Presence of any extra-hepatic metastases
* Presence of main portal vein (PV) or inferior vena cava (IVC) involvement
* Presence of active, uncontrolled varices
* Presence of active, severe comorbidities including uncontrolled cardiovascular or cerebrovascular diseases or recent events within 6months prior to treatment
* Received prior non-curative locoregional (including TACE, RT to liver, SIRT) or systemic therapy received for HCC\
* Prior treatment with any anti-programmed cell death protein-1 (anti-PD-1), PD Ligand-1 (PD-L1) or PD Ligand-2 (PD-L2) agent, or an antibody targeting other immune-regulatory receptor(s) or mechanism(s)
* Use of chronic systemic steroid or any other immunosuppressive medication within 14days prior to treatment initiation, except:
* Intranasal, inhaled, topical steroids, or local steroid injection;
* Systemic corticosteroids at physiologic doses ≤10mg/day of prednisone or equivalent;
* Steroids as premedication for hypersensitivity reactions
* Active or documented autoimmune or inflammatory disorders within 2years, except diabetes type I, vitiligo, psoriasis, or hypo-/hyperthyroid diseases not requiring immunosuppressant(s)
* Known history of a positive HIV test, primary/acquired immunodeficiency syndrome, or solid organ transplantation
* Receipt of live, attenuated vaccine within 28 days prior to study treatment
* Severe hypersensitivity reaction to another monoclonal antibody
* Presence of any contraindication to TACE not otherwise listed: cisplatin allergy
* Presence of any contraindication to SBRT not otherwise listed:
* Maximal size of any one HCC >25 cm
* Direct tumour extension into gastrointestinal structures (stomach, duodenum, remaining small or large bowel)
* Presence of any contraindication to SIRT not otherwise listed:
* Pre-treatment 99mTc-MAA scan >20% lung shunting of hepatic artery blood flow, or a demonstration of radiation exposure to the lungs potentially >25Gy
* Pre-treatment hepatic angiogram showing potential Y90 microspheres deposition in the gastrointestinal tract or any other organ(s) which is not correctable by catheter embolization techniques.
* Pregnant or lactating females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2034-03-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | defined as the period from the date of starting TACE or Y90-radioembolisation to the time of local, in-field disease progression, or the time of patient death, whichever occurring first; up to 10 years

SECONDARY OUTCOMES:
Overall Survival (OS) | defined as the period from the date of starting TACE or Y90-radioembolisation to the date of patient death; up to 10 years
Objective response rate (ORR) per mRECIST criteria | The percentage of patients in each study group achieving a partial response or complete response to intervention arm, from start of TACE or SIRT to date of progression or death; up to 10 years
  treatment response measurement
Local Control (LC) | From start of TACE or SIRT to local (target lesion) progression or death, whichever occurs first; up to 10 years
  Defined as the absence of progressive disease within the PTV per mRECIST, i.e. the sum of Clinical Remission (CR), Partial Response (PR) and Stable Disease (SD)
Surgical conversion rate | From treatment to disease progression or death, up to 10 years
  Defined as the percentage of patients amendable to curative surgical interventions or transplantation after successful tumour(s) down-sizing by intervention treatment
Pathological response | From treatment completion to disease progression or death; up to 10 years
  Defined as the percentage of surface with non-viable cancer cells (represented by necrosis or fibrosis) in relation to the total tumour area = 100% - viable cancer cells (%).
Factors independently associated with survival outcomes of treated patients | From start of treatment to progression or death of treated patients; up to 10 years
  Baseline characteristics are to be recorded and analyzed using univariate and multivariate analyses to identify factors independently associated with survival outcomes of treated patients
Safety outcome measures | From start of treatment to progression or death of treated patients; up to 10 years
  Incidence, nature, and severity of adverse events graded according to the United States National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE 5.0)
Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) questionnaire | From pre-treatment baseline to disease progression or death; up to 10 years
  To assess patient-reported quality of life by means of serial FACT-Hep validated questionnaire; the score ranges from 0-180, with a higher score representing a better quality of life.
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core-30 (QLQ-C30) Questionnaire | From pre-treatment baseline to disease progression or death; up to 10 years
  To assess patient-reported quality of life by means of serial European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core-30 (QLQ-C30) validated questionnaire. The EORTC QLQ-C30 scale score ranges from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptomatology.
Radiomics | From pre-treatment baseline imaging to the last imaging before the death of treated patients; for up to 10 years
  To develop a radiomics model with robust features for survival prediction of liver cancer patient after SIRT or SBRT; through analysis of diagnostic and progress CT imaging features in study participants
Predictive Biomarkers | From pre-treatment baseline blood tests to the last before the death of treated patients; for up to 10 years
  Potential, predictive blood biomarkers, including peripheral mononuclear cells (PBMC), exosomal PD-L1 are serially measured during individual patients' entire treatment course

CONTACTS AND LOCATIONS:
Locations (1):
- Tuen Mun Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Wong N, Chiang C, Ho C, Yip W, Yeung C, Chan M, et al. Prognostic Factors and Survival in Advanced Large Hepatocellular Carcinomas Treated with Combined Transarterial Chemoembolisation and Hypofractionated Image-guided Radiotherapy. Hong Kong Journal of Radiology. 2020 Sep 25;23(3):198-207.
- [Background] Chiang CL, Chan KSK, Chiu KWH, Lee FAS, Chen W, Wong NSM, Ho RLM, Lee VWY, Man K, Kong FMS, Chan ACY. Complete Response to Locoregional Therapy Plus Immunotherapy for Hepatocellular Carcinoma. JAMA Oncol. 2024 Nov 1;10(11):1548-1553. doi: 10.1001/jamaoncol.2024.4085. PMID 39325464
- [Background] Chiang CL, Lee FAS, Chan KSK, Lee VWY, Chiu KWH, Ho RLM, Fong JKS, Wong NSM, Yip WWL, Yeung CSY, Lau VWH, Man K, Kong FMS, Chan ACY. Survival Outcome Analysis of Stereotactic Body Radiotherapy and Immunotherapy (SBRT-IO) versus SBRT-Alone in Unresectable Hepatocellular Carcinoma. Liver Cancer. 2023 Oct 1;13(3):265-276. doi: 10.1159/000533425. eCollection 2024 Jun. PMID 38756147
- [Background] Chiang CL, Chiu KWH, Chan KSK, Lee FAS, Li JCB, Wan CWS, Dai WC, Lam TC, Chen W, Wong NSM, Cheung ALY, Lee VWY, Lau VWH, El Helali A, Man K, Kong FMS, Lo CM, Chan AC. Sequential transarterial chemoembolisation and stereotactic body radiotherapy followed by immunotherapy as conversion therapy for patients with locally advanced, unresectable hepatocellular carcinoma (START-FIT): a single-arm, phase 2 trial. Lancet Gastroenterol Hepatol. 2023 Feb;8(2):169-178. doi: 10.1016/S2468-1253(22)00339-9. Epub 2022 Dec 15. PMID 36529152
- [Background] de la Torre-Alaez M, Matilla A, Varela M, Inarrairaegui M, Reig M, Lledo JL, Arenas JI, Lorente S, Testillano M, Marquez L, Da Fonseca L, Argemi J, Gomez-Martin C, Rodriguez-Fraile M, Bilbao JI, Sangro B. Nivolumab after selective internal radiation therapy for the treatment of hepatocellular carcinoma: a phase 2, single-arm study. J Immunother Cancer. 2022 Nov;10(11):e005457. doi: 10.1136/jitc-2022-005457. PMID 36450386
- [Background] Dawson LA, Winter K, Knox J, Zhu AX, Krishnan S, Guha C, et al. NRG/RTOG 1112: Randomized Phase III Study of Sorafenib vs. Stereotactic Body Radiation Therapy (SBRT) Followed by Sorafenib in Hepatocellular Carcinoma (HCC) (NCT01730937). Int J Radiat Oncol. 2022 Dec;114(5):1057.
- [Background] Apisarnthanarax S, Barry A, Cao M, Czito B, DeMatteo R, Drinane M, Hallemeier CL, Koay EJ, Lasley F, Meyer J, Owen D, Pursley J, Schaub SK, Smith G, Venepalli NK, Zibari G, Cardenes H. External Beam Radiation Therapy for Primary Liver Cancers: An ASTRO Clinical Practice Guideline. Pract Radiat Oncol. 2022 Jan-Feb;12(1):28-51. doi: 10.1016/j.prro.2021.09.004. Epub 2021 Oct 21. PMID 34688956
- [Background] Wong SS, Wong WH, Ngar DY, Ma VW, Cheung C, Lee FA. NTWC Guideline for Transarterial Radioembolization using Yttrium-90 Microspheres (Y90-TARE). Hong Kong; 2020 Sep. (1).
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338